CLINICAL TRIAL: NCT01892293
Title: A Phase I/IIa, Open Label, Multiple Site Clinical Trial Evaluating the Safety and Activity of Engineered Autologous T Cells Expressing an Affinity-enhanced TCR Specific for NY-ESO-1 and LAGE-1 in Patients With Relapsed or Progressive Disease in Multiple Myeloma
Brief Title: CT Antigen TCR-Engineered T Cells for Myeloma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Adaptimmune (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADP-0011-002
Record Dates: First submitted 2013-06-27; First posted 2013-07-04 (Estimated); Results first posted 2018-07-24 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Autologous stem cell transplantation; Received initial treatment previously
MeSH Terms: conditions — Multiple Myeloma | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Autologous genetically modified T cells (Experimental): Patients with a confirmed diagnosis of myeloma, with measurable disease, and who have received prior therapy for their myeloma that includes an IMiDs and a proteasome inhibitor and who have relapsed or progressive disease, will receive treatment with NY-ESO-1c259-modified T cells. An intended total dose of ≥0.1-1e10 total cells will be administered as a single infusion. A low dose infusion of 1e8 to < 1e9 will be allowed for patients if cells do not expand sufficiently to reach the target dose range.
  Interventions: Drug: Treatment with NY-ESO-1c259-modified T cells

INTERVENTIONS:
Drug: Treatment with NY-ESO-1c259-modified T cells — An intended total dose of ≥0.1-1e10 total cells will be administered as a single infusion. A low dose infusion of 1e8 to < 1e9 will be allowed for patients if cells do not expand sufficiently to reach the target dose range.
  For patients whose disease progresses and whose tumor still expresses tumor antigen and HLA-A201, a second infusion of up to 5e10 cells may be given.

SUMMARY:
This study will enroll patients with multiple myeloma who have received prior therapy for their disease but their disease has progressed or relapsed.

DETAILED DESCRIPTION:
The primary objective of the study is to evaluate the safety and tolerability of autologous genetically modified T cells transduced to express the high affinity NY-ESO-1c259 TCR in HLA-A201 patients. Eligibility screening will be performed in two steps. First, patients will undergo prescreening to determine if they have the correct HLA type in order to respond to the engineered T cell therapy, and to test for presence of the target antigen, NY-ESO-1 and LAGE-1, in their tumor cells. Patients, who are HLA-A201 positive and test positive for expression of NY-ESO-1 and/or LAGE-1 in their myeloma tumor will move on to complete all screening procedures to determine eligibility for the study.

Patients will initially undergo a steady-state mononuclear cell apheresis for T cell collection. About 3-4 weeks later (to allow expansion/engineering/releasing the engineered T cells), patients will receive a short course of cytoreductive chemotherapy prior to receiving the engineered T cell infusion, comprised of 1.5 gm/m2 of cyclophosphamide, mesna will be given if in accordance with institutional standards.

At day 0, patients will receive a dose of ≥0.1-1 x 1010 anti-CD3/anti-CD28-costimulated autologous T cells which have been genetically modified to express affinity-enhanced NY-ESO-1 T cell receptors (TCRs). A minimum dose of 0.1≤x<1 x 109 will be permitted. Patients receiving this low dose level will be evaluated separately for safety and efficacy.

Patients will undergo myeloma restaging approximately 1 week prior to the T cell infusion, and post infusion at days +28, +42 (week 6), +100 and 6 months post infusion and then every 3 months until relapse/progression or until 1 year, whenever comes first. At this point, patients will be followed semi-annually for up to 5 years and then annually for long term follow-up for monitoring for delayed adverse events until 15 years after receiving the genetically modified T cells, in accordance with FDA Guidelines.

ELIGIBILITY:
Inclusion Criteria:

* 1. Written informed consent must be obtained from all patients before entry into the study

  2. Patients must have a diagnosis of myeloma (see Appendix A for diagnostic criteria).

  3. Patients must have progressive or active disease following prior therapy for their myeloma which:
  1. includes an IMiD and proteasome inhibitor as separate lines or a combined line of therapy
  2. May include prior auto-SCT but not prior allo-SCT

     Patients who have failed second or third line therapy and beyond, such as DPACE, and who are experiencing a partial response rather than progressive disease are also eligible.

     4. Patients must have measurable disease on study entry. Measurable disease may include quantifiable or detectable levels of serum or urine paraprotein. For patients with minimally secretory disease on study entry, serum free kappa or lambda light chain levels, or the serum free light chain ratio may be measured and used for disease monitoring if abnormal.

     5. Patients must be HLA-A201 as determined by a CLIA certified (or equivalent) clinical laboratory. (This determination will be made under a pre-enrollment screening ICF)

     6. Patients must have confirmed expression of NY-ESO-1 and/or LAGE-1 by RT-PCR, immunohistochemistry or quantigene analysis. (This determination will be made under a pre-enrollment screening ICF)

     Exclusion Criteria:
* 1. Pregnant or nursing females 2. HIV or HTLV-1/2 seropositivity 3. Known history of myelodysplasia 4. Known history of chronic active hepatitis or liver cirrhosis (if suspected by laboratory studies, should be confirmed by liver biopsy).

  5. Active Infection with HBV or HCV
  * Active hepatitis B infection as determined by test for hepatitis B surface antigen.
  * Active hepatitis C. Patients will be screened for HCV antibody. If the HCV antibody is positive, a screening HCV RNA by any RT PCR or bDNA assay must be performed at screening by a local laboratory with a CLIA certification or its equivalent. Eligibility will be determined based on a negative screening value. The test is not required if documentation of a negative result of a HCV RNA test performed within 60 days prior to screening is provided.

    6. Prior allogeneic transplant 7. History of severe autoimmune disease requiring steroids or other immunosuppressive treatments.

    8. Active immune-mediated diseases including: connective tissue diseases, uveitis, sarcoidosis, inflammatory bowel disease, multiple sclerosis.

    9. Evidence or history of other significant cardiac, hepatic, renal, ophthalmologic, psychiatric, or gastrointestinal disease which would likely increase the risks of participating in the study. The specific type of stress test will be selected at the PI's discretion.

    10. Active bacterial or systemic viral or fungal infections.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-10-15 (Actual); Primary Completion 2014-12-10 (Actual); Study Completion 2018-04-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Stadtmauer, MD, Study Chair — University of Pennsylvania
Locations (2):
- United States (2):
  - City of Hope, Duarte, California
  - Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland

RESULTS

PARTICIPANT FLOW:
Groups:
- NY-ESO-1ᶜ²⁵⁹T Cells Administered IV: Participants who received cytoreductive chemotherapy followed by infusion of lentivirus-mediated genetically engineered NY-ESO-1ᶜ²⁵⁹T (Target dose: 1-10 billion cells)
Period: Overall Study
Arm/Group | NY-ESO-1ᶜ²⁵⁹T Cells Administered IV
Started | 6
Received T-cell | 2
Completed | 2
Not Completed | 4
Not completed — Apheresed but not treated | 4

BASELINE CHARACTERISTICS:
Population: Participants who received NY-ESO-1ᶜ²⁵⁹T
Arm/Group | NY-ESO-1ᶜ²⁵⁹T Cells Administered IV
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 1
Age, Continuous [Mean (Full Range); unit: Years] | 64.5 [61 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events Related to Study Treatment
Description: Number of Participants with NCI CTCAE Version 4.0 Adverse Events related to study treatment greater than or equal to Grade 3
Time Frame: Up to 12 months
Population: Participants who received NY-ESO-1ᶜ²⁵⁹T
Measure: Count of Participants; unit: Participants
Arm/Group | NY-ESO-1ᶜ²⁵⁹T Cells Administered IV
Number analyzed (Participants) | 2
Participants | 2

2. Secondary Outcome: Evaluate the Direct Anti-tumor Activity of NY-ESO-1ᶜ²⁵⁹T
Description: Number of participants with response post-infusion as assessed by international uniform response criteria
Time Frame: 180 days
Population: Participants who received NY-ESO-1ᶜ²⁵⁹T
Measure: Count of Participants; unit: Participants
Arm/Group | NY-ESO-1ᶜ²⁵⁹T Cells Administered IV
Number analyzed (Participants) | 2
Participants | 0

3. Secondary Outcome: Peak Persistence of Modified T-cells in the Peripheral Blood
Description: Measurement of NY-ESO-1ᶜ²⁵⁹T cells in blood (copies of WPRE per µg of genomic PBMC DNA)
Time Frame: Days 1, 3, 5, 8, 15, 22, 29, 43, 101, 130 181, every 3 months thereafter
Population: Participants who received cytoreductive chemotherapy followed by infusion of NY-ESO-1ᶜ²⁵⁹T with persistence data
Measure: Mean (Full Range); unit: copies per μg of DNA
Arm/Group | NY-ESO-1ᶜ²⁵⁹T Cells Administered IV
Number analyzed (Participants) | 2
copies per μg of DNA | 29,179 [4479 to 53,879]

ADVERSE EVENTS:
Time Frame: Start of lymphodepletion to end of intervention phase (up to 12 months post T-cell infusion)
Description: Participants who received NY-ESO-1ᶜ²⁵⁹T
Arm/Group | NY-ESO-1ᶜ²⁵⁹T Cells Administered IV
All-Cause Mortality (participants affected / at risk) | 2/2
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NY-ESO-1ᶜ²⁵⁹T Cells Administered IV (N=2)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NY-ESO-1ᶜ²⁵⁹T Cells Administered IV (N=2)
White blood cell count decreased (Investigations) | 2 (2)
Lymphocyte count decreased (Investigations) | 2 (2)
Neutrophil count decreased (Investigations) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Fatigue (General disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less